CLINICAL TRIAL: NCT05168306
Title: Evaluation of the Impact of the FreeStyle Libre 2 Flash Glucose Monitoring System, Compared to the Current Standard of Care (SOC), on Weight Reduction in Subjects With Type 2 Diabetes.
Brief Title: T2 FSL2 Weight Loss
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment and Study no longer required
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-RES-21215
Record Dates: First submitted 2021-12-20; First posted 2021-12-23 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: FreeStyle Libre
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Standard of Care: No intervention will be administered. Subjects randomized to the Standard of Care Arm will continue using their Current standard of care device to monitor and manage their diabetes
- Intervention: Subjects randomized to this Arm will use FreeStyle Libre 2 to monitor and manage their diabetes.
  Interventions: Device: FreeStyle Libre 2 Flash Glucose Monitoring System

INTERVENTIONS:
Device: FreeStyle Libre 2 Flash Glucose Monitoring System — The FreeStyle Libre 2 Flash Glucose Monitoring System is a continuous glucose monitoring (CGM) device with real time alarms capability indicated for the management of diabetes in persons age 4 and older.
  Groups: Intervention

SUMMARY:
To compare the impact of the FreeStyle Libre (FSL) 2 Flash Glucose Monitoring System to the current Diabetes Monitoring standard of care (SOC) on weight reduction in subjects with type 2 diabetes.

DETAILED DESCRIPTION:
This is a non-pivotal, randomized, two-arm, multi-center, prospective, non-significant risk study to evaluate the impact of the FreeStyle Libre 2 Flash Glucose Monitoring System compared to the current Diabetes Monitoring standard of care (SOC) on weight reduction in subjects with type 2 diabetes.

Subjects who have been diagnosed with type 2 diabetes will be randomized to use FreeStyle Libre 2 sensor (intervention arm) or their current standard of care (control arm) to manage their diabetes for a period of 6 months. Subjects will be asked to complete the Diabetes Treatment Satisfaction Questionnaire (DTSQ) at baseline (visit 1) and during visit 6. Subjects will also complete a separate subject questionnaire during visit 6.

All subjects will wear a FreeStyle Libre Pro sensor for enrollment (Screening) purposes and to collect baseline glycemic data prior to randomization. In addition, all subjects in both the intervention and control arms will wear an FSL Pro at days 75 and 165 for collection of glycemic endpoint data.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 30 years of age and no more than 70 years of age at the time of enrollment.
2. Subject must have laboratory-based HbA1c measurement of between 8.0% and 10.0%.
3. Subject has 25% or more time spent above 180 mg/dL between the hours of 6am and 10pm during the screening phase.
4. Subject has a Body Mass Index (BMI) of 30 or greater.
5. Subject must have had a diagnosis of type 2 diabetes.
6. Subject must be able to read and understand English and/or Spanish.
7. In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
8. Subject is willing to make diet and lifestyle changes in response to education and glucose data
9. Subject must be available to participate in all study visits.
10. Subject must be willing and able to provide written signed and dated informed consent.

    Exclusion Criteria:
11. Subject is unable to perform mild physical activity (i.e. walking, stationary bike, etc.) for a minimum of 20 minutes per day.
12. Subject has used an unblinded continuous glucose monitor in the three (3) months prior to enrollment.
13. Subject is currently on any form of insulin therapy.
14. Subject is currently on a low carbohydrate diet.
15. Subject is currently using a commercial structured-meal weight loss program (i.e. Nutrisystem)
16. Subject is currently taking sulfonylurea-based medications.
17. Subject has experienced weight loss or gain of 5% or more of their total weight within the past 90 days.
18. Subject is currently taking prescription weight loss drugs, including, but not limited to, bupropion-naltrexone (Contrave), liraglutide (Saxenda), orlistat (Xenical), phentermine-topiramate (Qsymia) and semaglutide (Wegovy).
19. Subject is currently taking over-the-counter medications or supplements purported to aid in weight loss.
20. Subject is currently taking intramuscular or intravenous corticosteroids.
21. Subject has previously undergone or is planning on undergoing gastric bypass, gastric banding or gastric sleeve surgery in the next six (6) months.
22. Subject is currently taking atypical antipsychotic medications.
23. Subject has a condition that can lead to development of secondary diabetes (including but not limited to cystic fibrosis, hemochromatosis, chronic pancreatitis, polycystic ovary syndrome (PCOS), Cushing's syndrome, having undergone a pancreatectomy).
24. Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
25. Subject is pregnant, attempting to conceive or not willing and able to practice birth control during the study duration (applicable to female subjects only).
26. Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. Such conditions include, but are not limited to extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, redness, infection or edema.
27. Subject is currently undergoing or is anticipated to undergo treatment for cancer (including but not limited to oral and/or intravenous chemotherapy, radiation treatment, surgery, bone marrow transplant).
28. Subject has untreated mental illness and/or opiate addiction.
29. Subject has concomitant medical condition which, in the opinion of the investigator, could present a risk to the safety or welfare of the subject or study staff.
30. Subject is currently undergoing dialysis and/or has end stage renal disease.
31. Subject is currently participating in another interventional clinical trial.
32. Subject is unsuitable for participation due to any other cause as determined by the investigator.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have been diagnosed with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-12-05 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Difference in bodyweight from the control arm at 6 months | six (6) months
  Subjects' bodyweight will be measured during Visits 1, 3, 5 and 7. At the end of the 6 months period the bodyweight change, if any, will be assessed between the two Arms of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara A Karinka, PhD, Study Director — Abbott Diabetes Care
Locations (1):
- Rainier Clinical Research Center, Renton, Washington, United States

IPD SHARING:
Plan to Share IPD: No